CLINICAL TRIAL: NCT01075334
Title: Is a Carnitine Based Food Supplement (PorimoreTM) for Infertile Men Superior to Folate and Zinc With Regard to Pregnancy Rates in Intrauterine Insemination Cycles?
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shaare Zedek Medical Center (Other)
Responsible Party: Avi Tsafrir, MD, IVF Unit, Shaare Zedek Medical Center, Jerusalem, Israel
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: porimore.CTIL
Record Dates: First submitted 2010-02-24; First posted 2010-02-25 (Estimated); Last update posted 2010-02-25 (Estimated); Status verified 2010-02

CONDITIONS: Male Infertility
Keywords: sperm; male infertility; Carnitine; food supplementation; insemination
MeSH Terms: conditions — Infertility, Male | interventions — Zinc

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Porimore arm (Experimental): Infertile men will receive 'Porimore' tablets for a period of time in which three intrauterine insemination cycles will be performed.
  Interventions: Dietary Supplement: Porimore - A Carnitine based food supplement
- Folate and Zinc (Active Comparator)
  Interventions: Dietary Supplement: Zinc and Folate Supplementation

INTERVENTIONS:
Dietary Supplement: Porimore - A Carnitine based food supplement — A daily dose of 2 grams L-carnitine, 1 gr acetyl L-carnitine, 500mg Vitamin C, 400 IU vitamin E, 60 mg Q10, 30mg Zinc Picolinate, 500mcg Folic Acid, 200 Mcg Selenium, 100 MCG Vitamin B12.
  Arms: Porimore arm
Dietary Supplement: Zinc and Folate Supplementation — 500 Mcg Folic acid, 30-60 mg Zinc tablets/ day
  Arms: Folate and Zinc

SUMMARY:
Many cases of male infertility are poorly understood and regarded as unexplained. Therefore, a etiological treatment for this condition can not be offered in most cases. A beneficial effect on sperm motility was found in trails using antioxidants such as carnitine, zinc and folic acid. However, most studies lacked a sufficient power to detect a significant effect on pregnancy rates. In this study, infertile men with abnormal sperm quality parameters will be randomized to receive either carnitine-based food supplement (Porimore) or folate and Zinc Tablets.

ELIGIBILITY:
Inclusion Criteria:

* infertility
* at least one abnormal sperm quality parameter
* female age < 35
* normal ovarian reserve

Exclusion Criteria:

* known allergy to one of the food additives planned for treatment

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2010-02; Primary Completion 2010-02 (Actual); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
Pregnancy Rate | 3 Insemination cycles
  proportion of women becoming pregnancy following treatment with intrauterine insemination

SECONDARY OUTCOMES:
Sperm quality parameters | 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- Shaare-Zedek IVF and infertility unit, Jerusalem, Israel

REFERENCES:
- [Background] Isidori AM, Pozza C, Gianfrilli D, Isidori A. Medical treatment to improve sperm quality. Reprod Biomed Online. 2006 Jun;12(6):704-14. doi: 10.1016/s1472-6483(10)61082-6. PMID 16792845
- [Derived] de Ligny W, Smits RM, Mackenzie-Proctor R, Jordan V, Fleischer K, de Bruin JP, Showell MG. Antioxidants for male subfertility. Cochrane Database Syst Rev. 2022 May 4;5(5):CD007411. doi: 10.1002/14651858.CD007411.pub5. PMID 35506389